CLINICAL TRIAL: NCT04958928
Title: A Prospective, Multicenter, Cohort Study of Termination of Persistent Atrial Fibrillation by Catheter Ablation
Brief Title: Termination of Persistent Atrial Fibrillation by Catheter Ablation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Wuhan Central Hospital (Other); Ruijin Hospital (Other); Beijing Chao Yang Hospital (Other); The Third Xiangya Hospital of Central South University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Xiamen Cardiovascular Hospital, Xiamen University (Other); The Third People's Hospital of Chengdu (Other)
Responsible Party: Principal Investigator, Xu Liu, Professor, Shanghai Chest Hospital
Other Study IDs: Termination-AF
Record Dates: First submitted 2021-07-06; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persistent AF Group
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Catheter ablation — All patients received radiofrequncy ablation.

SUMMARY:
This is a prospective, multicenter, cohort study aims to demonstrate the role of termination of AF in ablation for persistent atrial fibrillation, and evaluate the clinical outcomes in patients with or without AF termination.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years old; 2. Persistent AF; 3. Nonresponse or intolerance to ≥1 antiarrhythmic drug.

Exclusion Criteria:

1. With uncontrolled congestive heart failure;
2. Having significant valvular disease and/or prosthetic heart valve(s);
3. With myocardial infarction or stroke within 6 months of screening;
4. With Significant congenital heart disease;
5. Ejection fraction was <40% measured by echocardiography;
6. Allergic to contrast media;
7. Contraindication to anticoagulation medications;
8. Severe pulmonary disease e.g. restrictive pulmonary disease, chronic obstructive disease (COPD);
9. Left atrial (LA) thrombus measured by pre-procedure transesophageal echocardiography;
10. Having any contraindication to right or left sided heart catheterization; 11. Previous atrial fibrillation ablation;

12. Presence of an implanted cardioverter-defibrillator; 13. Any cardiac surgery within the past 2 months; 14. Poor general health; 15.Life expectancy less than 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent AF.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
AF recurrence rate | 12 months
  AF recurrence is defined as presence of documented AF episodes of 30 recurrence is defined as presence of documented AF episodes of 30 seconds or longer duration.

IPD SHARING:
Plan to Share IPD: Yes